CLINICAL TRIAL: NCT00839683
Title: Pharmacokinetic Drug Interaction Study of Dapagliflozin and Valsartan or Simvastatin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MB102-036
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Simvastatin; dapagliflozin; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- simvastatin (Active Comparator)
  Interventions: Drug: simvastatin
- Dapagliflozin + simvastatin (Active Comparator)
  Interventions: Drug: Dapagliflozin; Drug: simvastatin
- Dapagliflozin (Active Comparator)
  Interventions: Drug: Dapagliflozin
- valsartan (Active Comparator)
  Interventions: Drug: valsartan
- Dapagliflozin + valsartan (Active Comparator)
  Interventions: Drug: Dapagliflozin; Drug: valsartan

INTERVENTIONS:
Drug: simvastatin — Tablets, Oral, 20 mg, Single Dose
  Other Names: Zocor
  Arms: simvastatin
Drug: Dapagliflozin — Tablets, Oral, 20 mg, Single Dose
  Other Names: BMS-512148
  Arms: Dapagliflozin; Dapagliflozin + simvastatin; Dapagliflozin + valsartan
Drug: simvastatin — Oral, 40 mg, Single Dose
  Arms: Dapagliflozin + simvastatin
Drug: valsartan — Tablets, Oral, 320 mg, Single Dose
  Other Names: Diovan
  Arms: Dapagliflozin + valsartan; valsartan

SUMMARY:
Phase A - To assess the effect of simvastatin on the pharmacokinetics (PK) of dapagliflozin and to determine the effect of dapagliflozin on the PK of simvastatin, when simvastatin and dapagliflozin are coadministered in healthy subjects. Phase B - To assess the effect of valsartan on the PK of dapagliflozin and to determine the effect of dapagliflozin on the PK of valsartan, when valsartan and dapagliflozin are coadministered in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m2, inclusive. BMI = weight (kg)/[height (m)]2

Exclusion Criteria:

* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 12 weeks after the last dose of investigational product
* Abnormal urinalysis at screening (repeat urinalysis may be allowed for positive hematuria in women)
* Glucosuria at screening
* Abnormal liver functions tests (ALT, AST or total bilirubin > 10% above ULN)
* Presence of edema on physical exam
* History of diabetes mellitus
* History of heart failure
* History of renal insufficiency
* History of chronic or recurrent UTI (defined as 3 occurrences per year) or UTI in the past 3 months
* History of recurrent (defined as 3 occurences per year) or recent vulvovaginal mycotic infections
* Positive urine screen for drugs of abuse either at screening or before dosing
* Positive blood screen for hepatitis C antibody, hepatitis C antibody, hepatitis B surface antigen, or HIV-1, -2 antibody
* History of allergy to SGLT2 inhibitors or related compounds
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity)
* History of allergy or intolerance to valsartan or simvastatin (or related compounds)
* Prior exposure to dapagliflozin, valsartan or simvastatin within 3 months of Day -1
* Exposure to any investigational drug or placebo within 4 weeks of Day -1
* Use of any prescription drugs within 4 weeks or over-the-counter acid controllers within 2 weeks prior to any study drug administration
* Use of any other drugs, including over-the counter medications within 1 week and herbal preparations within 2 weeks prior to admission to the study facility
* Use of an oral, injectable or implantable hormonal contraceptive agent within 3 months of Day -1

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Exposure to the investigational drug will be measured to compare with and without the co-administration of other drugs | 72 hours post-dose

SECONDARY OUTCOMES:
To assess the safety and tolerability of dapagliflozin when administered alone, with valsartan, or with simvastatin in healthy subjects | 15 timepoints
To assess the safety and tolerability of the combination of dapagliflozin with valsartan, and the combination of dapagliflozin with simvastatin in healthy subjects | 15 timepoints
To assess the effect of dapagliflozin on the PK of simvastatin acid (active metabolite of simvastatin), when coadministered in healthy subjects | 15 timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Mds Pharma Services (Us) Inc., Neptune City, New Jersey, United States

REFERENCES:
- See also: MB102-036_redacted _CSR _synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3642&filename=MB102-036_redacted%20_CSR%20_synopsis.pdf